CLINICAL TRIAL: NCT06570525
Title: Improving Traumatic Stress in Women Who Have Experienced Homelessness: Evaluation of a Stakeholder Engaged Intervention
Brief Title: Intervention Evaluation WEH (Women Who Have Experienced Homelessness)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Principal Investigator left the institution
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24061301
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NurseNET-Narrative Exposure Therapy (Experimental): Nurse-Delivered Narrative Exposure Therapy (NurseNET). Narrative Exposure Therapy (NET) is a brief, low-cost, trauma-focused treatment modality that is effective in treating mobile populations with complex PTSD. In NurseNET, NET is facilitated by a clinically experienced nurse, while peers/program support specialists offer scaffolded support, fostering trust, engagement, and retention. NurseNET begins with administration of a "diagnostic battery" and psychoeducation. Then, in subsequent NurseNET sessions, using gradual imaginative exposure, the nurse guides the participant to verbally express and re-frame their personal trauma narratives to shift unhelpful beliefs/symptoms around trauma. NurseNET utilizes a racism-conscious approach to create relational spaces in which narratives of WEH are positioned to challenge dominant social narratives. Each NurseNET session offers a brief soulfulness-based stress reduction activity to prompt emotional/affective grounding.
  Interventions: Behavioral: NurseNET
- PAL: Peer Active Listening (Active Comparator): Peer Active Listening (PAL). In the PAL active comparator/control, peers/program support specialists meet individually with participants in "active listening sessions", along the same visit sequence as NurseNET. During PAL sessions, peers/program support specialists allow participants to set each conversational agenda while practicing the tenets of active listening, including attending to body language, paraphrasing the participant's verbal expressions, reflecting feelings, and using tactful repetition. PAL sessions are not intended to center on topics of trauma, but rather designed to offer a supportive relationship (attentional control).
  Interventions: Other: PAL

INTERVENTIONS:
Behavioral: NurseNET — Nurse-Delivered Narrative Exposure Therapy (NurseNET). Narrative Exposure Therapy (NET) is a brief, low-cost, trauma-focused treatment modality that is effective in treating mobile populations with complex PTSD. In NurseNET, NET is facilitated by a clinically experienced nurse, while peers/program support specialists offer scaffolded support, fostering trust, engagement, and retention. NurseNET begins with administration of a "diagnostic battery" and psychoeducation. Then, in subsequent NurseNET sessions, using gradual imaginative exposure, the nurse guides the participant to verbally express and re-frame their personal trauma narratives to shift unhelpful beliefs/symptoms around trauma. NurseNET utilizes a racism-conscious approach to create relational spaces in which narratives of WEH are positioned to challenge dominant social narratives. Each NurseNET session offers a brief soulfulness-based stress reduction activity to prompt emotional/affective grounding.
  Arms: NurseNET-Narrative Exposure Therapy
Other: PAL — Peer Active Listening (PAL). In the PAL active comparator/control, peers/program support specialists meet individually with participants in "active listening sessions", along the same visit sequence as NurseNET. During PAL sessions, peers/program support specialists allow participants to set each conversational agenda while practicing the tenets of active listening, including attending to body language, paraphrasing the participant's verbal expressions, reflecting feelings, and using tactful repetition. PAL sessions are not intended to center on topics of trauma, but rather designed to offer a supportive relationship (attentional control).
  Arms: PAL: Peer Active Listening

SUMMARY:
Homelessness and associated traumas disproportionately impact women relative to men. Women who have experienced homelessness (WEH) universally face traumatic stress, often before becoming homeless and while experiencing homelessness.

For WEH who are incarcerated, additional trauma may occur while in correctional settings. Black WEH are disproportionately impacted by trauma, homelessness, and incarceration, as is related to structural and individual racism and discrimination (racial trauma).

DETAILED DESCRIPTION:
Homelessness and associated traumas disproportionately impact women relative to men. Women who have experienced homelessness (WEH) universally face traumatic stress, often before becoming homeless and while experiencing homelessness. For WEH who are incarcerated, additional trauma may occur while in correctional settings. Black WEH are disproportionately impacted by trauma, homelessness, and incarceration, as is related to structural and individual racism and discrimination (racial trauma). In our stepwise, multi-year research process, across hundreds of interviews, WEH identified trauma as their priority health issue. In response to a dearth of culturally acceptable trauma care models, our team pilot tested Narrative Exposure Therapy (NET)-a brief, human rights-informed treatment for complex PTSD in resource-limited settings. In this randomized controlled trial (RCT), we seek to understand whether supplementing nurse-delivered NET with peer/program support will strengthen its effects on PTSD, co-occurring symptoms, and social determinants of health outcomes compared to an attentional control, while optimizing implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* self-identifies as a woman
* ≥18 years of age
* history of homelessness or currently experiencing homelessness (HRSA criteria)
* affected by trauma-related distress (≥1 on Life Events Checklist + PTSD Checklist for DSM-5 ≥28)
* at least 75% of the sample must self-identify as Black/African American

Exclusion Criteria:

• impaired decisional capacity (UC-San Diego Brief Assessment ≤14.5)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder (PTSD) symptoms | Eligibility Screening; Pre-/Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5). Higher score = worse outcome. Range: 0-80.

SECONDARY OUTCOMES:
Depressive symptoms | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Patient Depression Questionnaire (PHQ-9). Higher score = worse outcome. Range: 0-27.
Anxiety | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Generalized Anxiety Disorder (GAD-7). Higher score = worse outcome. Range: 0-21.
Sleep symptoms | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Regensburg Insomnia Scale (RIS). Higher score = worse outcome. Range: 0-40.
Somatization | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Somatic Symptoms Scale (SSS-8). Higher score = worse outcome. Range: 0-32.
Substance use | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) tool. TAPS-1, is a four-item screening that asks about substance use in the past 12 months.

OTHER OUTCOMES:
Healthcare access | Pre-Assessment (week 0), Post-Assessment (week 4)
  Barriers to Access to Care Evaluation Scale (BACE). Higher score = worse outcome (greater barrier to seeking treatment). Range: 0-90. 30-items, 12-item subscale measures the extent to which stigma and discrimination are barriers to care.
Perceived social support | Pre-Assessment (week 0), Post-Assessment (week 4); Follow-up Assessments (weeks 10 and 16)
  Multidimensional Scale of Perceived Social Support Scale (MSPSS). Higher score = better. Range: 0-60.
Discrimination | Pre-Assessment (week 0), Post-Assessment (week 4)
  Everyday/Major Experiences of Discrimination Scale (EDS/MDS). This measure contains nine elements that assess the participant's perception of major experiences of discrimination, followed by a follow-up question about what the person believes was the reason for that discrimination (no numeric scoring).
Racial trauma | Pre-Assessment (week 0), Post-Assessment (week 4)
  Racial Trauma Scale (RTS) (short form research version). Higher score = worse. Range: 9-36.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten A Dickins, PhD, FNP-C, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No